CLINICAL TRIAL: NCT06014177
Title: A Digital Patient Decision Aid to Increase Sexually Transmitted Infection Testing in the Emergency Department: The STIckER Study
Acronym: STIckER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Jason E. Zucker, Assistant Professor of Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AAAU7485; 5R21AI168958 (NIH)
Record Dates: First submitted 2023-08-21; First posted 2023-08-28 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: STI; Sexually Transmitted Infection (STI); Sexually Transmitted Disease (STD)
Keywords: Gonorrhea; Chlamydia
MeSH Terms: conditions — Sexually Transmitted Diseases; Gonorrhea; Chlamydia Infections

STUDY DESIGN:
Intervention Model Description: Individuals will be randomized into the control arm (standard of care) or STIckER arm to receive the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): After enrollment but before the start of their clinical visit, participants assigned to a provider in the control arm will scan a QR code. They will receive a prompt stating, "If you would like to be tested for a sexually transmitted infection today, please tell your medical doctor."
  At the end of the visit, the participant will complete the "Patient Control Exit Survey" while the provider will complete the "Provider Control Exit Survey".
  These participants will not receive STIckER training.
  Interventions: Other: Control
- STIckER (Experimental): After enrollment but before the start of their clinical visit, participants assigned to a provider in the intervention arm will scan a QR code using their personal mobile phone at the start of their ED visit. If they do not have a mobile phone present, a secure password-protected tablet will be provided by the research staff. This will lead them to go through the STIckER decision aid modules. After completing the modules, participants will show the final outcome to their ED provider which may facilitate an SDM conversation about STI testing.
  At the end of the visit, the participant will complete the "Patient Intervention Exit Survey" while the provider will complete the "Provider Intervention Exit Survey.
  Interventions: Behavioral: STIckER

INTERVENTIONS:
Behavioral: STIckER — STIckER is an interactive and personalized intervention based on the principles of SDM that has been designed with input from the AYA ED patients and providers. STIckER guides AYA patients through a series of steps, beginning with "scanning your STIckER." Participants complete risk assessments, SDM modules, and conclude with an anonymous final digital infographic that informs an SDM conversation with the medical provider. This decision aid seamlessly integrates into the ED workflow, recommending appropriate STI testing for high-risk individuals and using SDM concepts for those at intermediate risk.
  Arms: STIckER
Other: Control — After enrollment but before the start of their clinical visit, AYA participants assigned to a provider in the control arm will scan a QR code. They will receive a prompt stating, "If you would like to be tested for a sexually transmitted infection today, please tell your medical doctor."
  Arms: Control

SUMMARY:
This study is a pilot randomized trial of STIckER in which 40 providers (20 trained in using the STIckER decision aid and 20 providing standard care) will enroll a total of 140 sexually active young Emergency Department (ED) patients over six months in a pediatric and adult ED setting. The primary goal is to determine if sexually active young individuals who use STIckER are more likely to undergo STI testing. By developing an effective automated digital tool to increase STI testing, the investigators aim to improve evidence-based sexual health education, reduce STI rates, and enhance the health outcomes of young individuals nationwide.

DETAILED DESCRIPTION:
Improving sexually transmitted infection (STI) screening is vital to combat the STI epidemic, especially among adolescents and young adults (AYA) aged 15-24 years in the United States. Inadequate testing for STIs in different body areas contributes to disease transmission. Emergency Departments (EDs) treat a significant number of young individuals, many of whom come from economically disadvantaged backgrounds and minority communities. Previous research has shown inconsistent use of contraception in this population, and despite the willingness of ED providers to support sexual health interventions, time and resource limitations present implementation challenges. To address this issue, the investigators propose developing STIckER (STI ChecK in the ER), a digital patient decision aid for STI testing in the ED that promotes shared decision-making. STIckER involves three steps: (1) patients complete a nonjudgmental sexual health screening assessment by scanning a quick-response (QR) code, (2) educational modules facilitate shared decision-making (SDM) by connecting personalized STI risk with evidence-based testing recommendations, and (3) a confidential, color-coded digital infographic aids the patient-provider discussion on STI testing.

ELIGIBILITY:
Inclusion Criteria:

* AYA aged 14-24 years
* Sexually active within the past 6 months (per self-report)
* Ability to speak English

Exclusion criteria:

* Severe illness
* Cognitive impairment
* Inability to speak English

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 184 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-06-13 (Actual)

PRIMARY OUTCOMES:
ED STI Testing Rate | Day 0
  Percent of individuals with any gonorrhea or chlamydia testing performed in the ED on the day of their STIckER visit.

SECONDARY OUTCOMES:
Extragenital STI testing Rate | Day 0
  Percent of individuals with any gonorrhea or chlamydia extra-genital (pharyngeal or rectal) test performed in the ED on the day of their STIckER visit.
Genitourinary STI testing Rate | Day 0
  Percent of individuals with any gonorrhea or chlamydia genitourinary test performed in the ED on the day of their STIckER visit.
STI Positivity Rate | Day 0
  Percent of individuals testing positive for gonorrhea or chlamydia at any site.
Acceptability of Intervention Measure (AIM) Score | At completion of all patient visits (within 6 months of enrollment)
  Acceptability assessed by a four item questionnaire with each question scored from 1 (completely disagree) to 5 (completely agree). Scores to each question are averaged to determine a mean score, ranging from 1 (minimum) to 5 (maximum), with a higher score indicating a better outcome.
Intervention Appropriateness Measure (IAM) Score | At completion of all patient visits (within 6 months of enrollment)
  Appropriateness assessed by a four item questionnaire with each question scored from 1 (completely disagree) to 5 (completely agree). Scores to each question are averaged to determine a mean score, ranging from 1 (minimum) to 5 (maximum), with a higher score indicating a better outcome.
Feasibility of Intervention Measure (FIM) Score | At completion of all patient visits (within 6 months of enrollment)
  Feasibility assessed by a four item questionnaire with each question scored from 1 (completely disagree) to 5 (completely agree). Scores to each question are averaged to determine a mean score, ranging from 1 (minimum) to 5 (maximum), with a higher score indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Zucker, MD, Principal Investigator — Columbia University; Lauren Chernick, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Children's Hospital of New York (CHONY), New York, New York
  - Milstein Hospital at NewYork-Presbyterian Hospital /Columbia University Irving Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No